CLINICAL TRIAL: NCT06421415
Title: Long Term Effect of AIT in Children
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HCA-AIT
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Allergy in Children
MeSH Terms: interventions — Desensitization, Immunologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Allergen Immunotherapy Extract — Patients will be treated as usual. The study is an observation of the long term effect of the treatment

SUMMARY:
The present study will investigate the long term effect of allergen immunotherapy in a real-life study in children with allergy undergoing subcutaneous or sublingual immunotherapy with grass pollen, birch, house dust mites or venom.

DETAILED DESCRIPTION:
The study will include children aged 5- 18 years who are treated with immunotherapy at Hans Christian Andersen Children' Hospital, Odense University Hospital.

Informed consent to be registered in a database and to receive a questionnaire 5 and 10 years after end of treatment are obtained before start of immunotherapy.

Base line data include information from the patient record: symptoms, medication, blood test and skin prick test results. During treatment effect, medication use, lung function and adverse events are monitored systematically once a year.

The questionnaires 5 and 10 years after end of treatment will focus on allergy symptoms, use of medication and asthma symptoms.

ELIGIBILITY:
Inclusion Criteria: treated with allergen immunotherapy at HCA Children'sHospital, Odense University Hospital -

Exclusion Criteria: received less than 12 months of treatment with allergen immunotherapy

-

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with moderate to severe allergy to grass pollen, birch, house dust mites or venom who are prescribed allergen immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2036-12-01 (Estimated); Study Completion 2037-05-01 (Estimated)

PRIMARY OUTCOMES:
Effect of immunotherapy 5 years after end of treatment | 5 years
  Medication use for allergy and asthma and the patient's experience of effect of the AIT on a scale from 0-4 (0= no effect, 1= modest effect, 2= some effect, 3= good effect, 4= very good effect)

SECONDARY OUTCOMES:
Effect of immunotherapy 10 years after end of treatment | 10 years
  Medication use for allergy and asthma and the patient's experience of effect of the AIT on a scale from 0-4 (0= no effect, 1= modest effect, 2= some effect, 3= good effect, 4= very good effect)

CONTACTS AND LOCATIONS:
Overall Officials: Josefine Gradman, PhD, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Hans Christian Andersen Children's Hospital, Odense, Odense C
  - Hans Christian Andersen Children's Hospital, Odense

IPD SHARING:
Plan to Share IPD: No